CLINICAL TRIAL: NCT04366414
Title: Breathing Protocol on Oxygen Saturation Recovery After a Dynamic Apnoea in Breath-hold Divers: a Single-blind, Randomized Clinical Trial
Brief Title: Breathing Protocol in Breath-hold Divers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Fran de Asís Fernández, Principal Investigator, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSEULS-PI-215/2018
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Exercise Training; Apnea; Breathholding; Breathing Exercises
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Intervention Model Description: parallel-group
Who Masked: Outcomes Assessor
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hook breathing removing nose-clip (Active Comparator): It will apply a usual training program for 4 weeks, 4hours and 30 min per week distributed equally over 3 days in the week. In each session, it was performed 8 submaximes-dynamic apnoeas with 3-minute recovery between each one. Then was performed a maximal-dynamic apnoea. To finish the session, was performed a continuous training of free style swimming at moderate effort over 30 minutes.
  During that training, only this group will perform an experimental breathing protocol consisted of removing nose-clip previous to surface and then perform hook breathing during 20 seconds. This protocol was applied at the end of each of the 8 submaximes-dynamic apnoeas and after the maximal-dynamic apnoea
  Interventions: Other: hook breathing removing nose-clip
- usual breathing (UB) (Active Comparator): It will apply a usual training program for 4 weeks, 4hours and 30 min per week distributed equally over 3 days in the week. In each session, it was performed 8 submaximes-dynamic apnoeas with 3-minute recovery between each one. Then was performed a maximal-dynamic apnoea. To finish the session, was performed a continuous training of free style swimming at moderate effort over 30 minutes.
  Interventions: Other: usual breathing (UB)

INTERVENTIONS:
Other: hook breathing removing nose-clip — Participants will perform 3 days per week of usual training, involving intense exercise 8 submaximes-dynamic apnoeas with 3-minute recovery between each one per session, and continuous training of free style swimming at moderate effort over 30 minutes, including warm-up, recovery between intervals and cool down.
  The experimental breathing protocol consisted on to remove nose-clip previous to surface and then perform hook breathing during 20 seconds.
  Arms: hook breathing removing nose-clip
Other: usual breathing (UB) — Participants will perform 3 days per week of usual training, involving intense exercise 8 submaximes-dynamic apnoeas with 3-minute recovery between each one per session, and continuous training of free style swimming at moderate effort over 30 minutes, including warm-up, recovery between intervals and cool down.
  Arms: usual breathing (UB)

SUMMARY:
The aim of this randomized controlled trial study was to assess the effects of an 4-week exercise program on the recovery capacity after a voluntary maximal apnea. Participants will be randomly allocated to perform an experimental breathing protocol (NR-HB), or an usual training using their usual breathing (UB) protocol.

DETAILED DESCRIPTION:
It is a multi-center study. 2 different Spanish Freedivers Centres are included in the study (Madrid and Zaragoza).

Divers were randomly assigned to receive an experimental training (NR-HB) or to be included in the Control Group (UB).

The trial included two study visits. Each exercise training program will be applied sessions per week during 4 weeks. Participants received baseline assessments at the beginning of any intervention, and post-intervention assessments at the end of the fourth week.

ELIGIBILITY:
Inclusion Criteria:

* Absence of pain or illness
* No changes in cognitive ability
* Over 18 years old.
* Member of the Spanish Federation of Underwater Activities.
* Positive medical examination that allows the diver to practice voluntary apnea.

Exclusion Criteria:

* People with systemic diseases, tumors, infections, pacemakers, history of epilepsy, hydrophobia, pregnancy women, pharmacological treatment.
* To be participating in other physical activities during the experimental research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-14 (Estimated)

PRIMARY OUTCOMES:
Oxygen Saturation change | Before and after training intervention (after 4 weeks)
  Oxygen Saturation recovery will be record by the experimenters every 5 seconds by a handheld pulse-oximeter during the 1 min recovery time after a maximal dynamic apnea. The outcome was the length of the time to return to 95% SpO2 during the 1 min recovery time after maximal dynamic apnoea

SECONDARY OUTCOMES:
Heart Rate recovery | before and after training intervention (after 4 weeks)
  Heart Rate will be record by the experimenters every 5 seconds by a handheld pulse-oximeter during the 1 min recovery time after a maximal dynamic apnea. The outcome was the length of the time to stabilize heart rate during these 1 minute.
Lung function (forced spirometry) | before and after training intervention (after 4 weeks)
  The Spirometry will be perform according to American Thoracic Society criteria and was measured in litres. The maneuver will be perform 3 times and recording the best one.

CONTACTS AND LOCATIONS:
Locations (1):
- Madrid FREEDIVERS association, Madrid, Spain

REFERENCES:
- [Background] Andersson JP, Liner MH, Runow E, Schagatay EK. Diving response and arterial oxygen saturation during apnea and exercise in breath-hold divers. J Appl Physiol (1985). 2002 Sep;93(3):882-6. doi: 10.1152/japplphysiol.00863.2001. PMID 12183481